CLINICAL TRIAL: NCT06722469
Title: A Randomized Controlled Trial Evaluating a Mobile Messenger-initiated, Theory-based, Culturally Tailored, and Fully Automated Chatbot to Increase Breast Cancer Screening Uptake
Brief Title: A Randomized Controlled Trial to Increase Breast Cancer Screening Uptake
Acronym: BCS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Thomas Yuen Tung Lam, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2024.527
Record Dates: First submitted 2024-11-21; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer Prevention; Breast Cancer Risk
Keywords: breast cancer; automated chatbot; breast cancer screening; health belief model
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either join the whatsapp chatbot intervention and standard text reminder group.
Who Masked: Participant
Masking Description: Participants will not know what arm they are randomized into.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- WCI (Experimental): The WCI group will receive automated messages based on the Health Belief Model (HBM) and Protection Motivation Theory (PMT), including personalized risk assessments, educational videos featuring medical professionals and relatable scenarios, and tailored prompts to encourage mammographic screening.
  Interventions: Other: WCI
- STR (No Intervention): A standard tet reminder will be sent regarding the breast cancer screening program

INTERVENTIONS:
Other: WCI — The WCI group will receive automated messages based on the Health Belief Model (HBM) and Protection Motivation Theory (PMT), including personalized risk assessments, educational videos featuring medical professionals and relatable scenarios, and tailored prompts to encourage mammographic screening.
  Arms: WCI

SUMMARY:
Breast cancer (BC) is the fifth leading cause of cancer deaths in women worldwide. In Hong Kong (HK), BC is the most common cancer, ranking third in cancer deaths among females. International guidelines advocate regular mammographic screening for women aged 40-50 to 69-74, reducing BC mortality by 20%.

The success and effectiveness of an organized cancer screening program are largely dependent on high adherence or uptake rates. However, nonadherence to BC screening is common and the suboptimal uptake rate remains a challenge, particularly in Asian countries.

Conventional interventions are effective in increasing mammographic screening uptake but are time-consuming, labor-dependent, and expensive. Mobile messenger chatbots are a potential cost-saving tool for enhancing BC screening uptake because they involve only a one-off development cost and a small maintenance cost . Currently, most studies evaluating the effectiveness of mobile health interventions in improving mammography screening uptake have been conducted in Western populations . Health-seeking behaviors for cancer screening in the Chinese population differ from those of Caucasians because of differences in culture, health beliefs, and education, especially regarding breast-related diseases. Chinese women often feel embarrassed when talking with healthcare workers in person about breast health. Communicating with a fully automated chatbot can minimize embarrassment. Additionally, linguistically and culturally tailored interventions are effective in increasing cancer screening rates in the Chinese population.

However, studies evaluating combined theory-based mHealth interventions to enhance BC screening uptake are scarce. Two theory-based WhatsApp chatbots were developed to promote CRC screening, and the longitudinal repeat fecal immunochemical test (FIT) adherence rate of a population-based CRC screening program in HK. These two chatbots used in investigator's previous studies had designs similar to that of the proposed chatbot, except for the health education materials. The chatbot design can be adopted directly with minor modifications to the workflow, replacement of content from CRC screening-related to BC screening-related, and culturally modified education materials. Consequently, the investigators can develop a new chatbot for this study at a lower cost and in a shorter time.

DETAILED DESCRIPTION:
In the past two decades, internet and mobile phone usage has increased due to affordability. The COVID-19 pandemic has further necessitated online and phone-based healthcare, paving the way for less labor-intensive, cost-effective mHealth interventions. These include short message service (SMS) text messages, telephone calls, email, social media, and mobile apps, which have significantly boosted BC screening uptake by 1.2%-50.9%. Among them, manual calls and SMS are prevalent methods. Manual calls facilitate interactions with subjects, aiding informed decision-making and participation but require high manpower. Although SMS offers automatic communication and chatbot features, each message costs approximately HKD$0.2, posing long-term economic challenges, especially for population-based interventions. Conversely, chatbots based on mobile messengers, like WhatsApp are less expensive due to unlimited free text and multimedia messaging across different mHealth operating systems. WhatsApp is globally prevalent, including in HK and has been successfully implemented in various clinical settings. Given these promising results, the investigators believe that mobile messenger-initiated chatbots have an extended role in the BC screening uptake rate because of the ubiquity, acceptability, and effectiveness of mHealth interventions. However, studies evaluating combined theory-based mHealth interventions to enhance BC screening uptake are scarce.

ELIGIBILITY:
Inclusion Criteria:

1. asymptomatic Chinese Women
2. 44-69 years old
3. eligible to enroll in a government-subsidized risk-stratified BC screening program
4. ability to read Chinese

Exclusion Criteria:

1. moderate- or high-risk women as defined by the local risk-stratified BC screening program
2. inability to provide informed consent
3. incomplete conversation with the chatbot.

Ages: 44 Years to 69 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — female
Enrollment: 470 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
BCS uptake rate | Within three months after the intervention
  The primary outcome is the BC screening uptake rate, defined as participation in and completion of mammographic screening within three months after the intervention.

SECONDARY OUTCOMES:
BCS uptake rate | Six months after the intervention
  BC screening uptake rate within six months after the intervention
Risk factors related to BCS non-adherence by interview | Six months after the intervention
  Risk factors associated with breast cancer screening non-adherence will be collected by focused group discussion
Mammography results | Six months after the intervention
  Number of positive mammography results of subjects who completed mammography
Mammograph breast biopsy rate | Six months after the intervention
  Uptake rate of subsequent breast biopsy for those with positive mammographic results
Detection rate of breast cancer | Six months after the intervention
  Detection rate of breast cancer

IPD SHARING:
Plan to Share IPD: Undecided
Still being decided